CLINICAL TRIAL: NCT03473158
Title: Early Fetal Reduction Through a Transvaginal Ultrasound Guided Approach in Multifetal Pregnancies: Mechanical Disruption Against Potassium Chloride Injection. A Randomized Controlled Trial
Brief Title: Fetal Reduction: Mechanical vs Chemical
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Riyadh Fertility and Reproductive Health center (Other)
Responsible Party: Principal Investigator, Ahmed AA Wali, MD, Lecturer of Obstetrics and Gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IVF-001-2018
Record Dates: First submitted 2018-03-09; First posted 2018-03-22 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Multiple Pregnancy
Keywords: fetal reduction; embryo reduction; feticide; potassium chloride; multiple pregnancy; multifetal pregnancy
MeSH Terms: interventions — Mechanical Thrombolysis; Potassium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical (Active Comparator): fetal reduction will be achieved by mechanical disruption of the fetal heart till asystole is achieved, and may be aided by partial or total suction of the fetus, using suction device attached to the embryo reduction needle
  Interventions: Device: Transvaginal ultrasound; Procedure: Mechanical fetal reduction
- Chemical (Active Comparator): fetal reduction will be achieved by injecting 0.5 mL of potassium chloride (Potassium Chloride® 15% , EIPICO, Egypt) into the cardiac region through the embryo reduction needle
  Interventions: Device: Transvaginal ultrasound; Procedure: Chemical fetal reduction

INTERVENTIONS:
Device: Transvaginal ultrasound — using the 6.5mHz intra-cavitary probe (65EC10EA) of ultrasound machine DP-50 (Shenzhen Mindray Bio-Medical Electronics Co., Ltd., P.R.China) to determine the number, site, size and cardiac activity of the fetuses, and monitor the fetal reduction procedure
Procedure: Mechanical fetal reduction — under transvaginal ultrasound guidance, fetal reduction will be achieved by mechanical disruption of the fetal heart till asystole is achieved, and may be aided by partial or total suction of the fetus, using suction device attached to the embryo reduction needle (Cook® Ireland Ltd., Limerick, Ireland)
  Other Names: Mechanical disruption
  Arms: Mechanical
Procedure: Chemical fetal reduction — under transvaginal ultrasound guidance, fetal reduction will be achieved by injecting 0.5 mL of potassium chloride (Potassium Chloride® 15% , EIPICO, Egypt) into the cardiac region through the embryo reduction needle (Cook® Ireland Ltd., Limerick, Ireland)
  Other Names: Potassium Chloride
  Arms: Chemical

SUMMARY:
In this study multifetal pregnancy reduction (to twins) will be carried out through a transvaginal route, at an early gestational age (6 weeks - 9weeks + 6days) using 2 methods: mere mechanical disruption against potassium chloride injection. The 2 methods will be compared regarding the efficacy, complications and pregnancy outcome.

DETAILED DESCRIPTION:
The incidence of multifetal gestations has increased dramatically over the past several decades. Multiple pregnancies are frequently complicated by maternal and fetal morbidities and mortalities. Data show that the incidence of morbidity and mortality correlate with fetal number. In the United Kingdom, the single embryo transfer policy has reduced the incidence of multifetal gestation. Also, in the United States the ASRM (American society of reproductive medicine) has revised the guidelines to optimize the number of transferred embryos during IVF. However in Egypt, transfer of 3 to 4 embryos is still practiced. The procedure of fetal reduction aims to decrease the occurrence of maternal and perinatal morbidities related to multifetal gestations. It can be carried out transvaginally or transabdominally under ultrasound guidance. It may be done by potassium chloride injection through needle injection, mere mechanical disruption by a needle, or by radiofrequency ablation. In this study multifetal pregnancy reduction will be carried out through transvaginal route, at an early gestational age (6 weeks - 9weeks + 6days), and compare the efficacy, complications and pregnancy outcome using mere mechanical disruption against potassium chloride injection.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with multifetal pregnancy (3 fetuses or more)
* Pregnant women from 6 weeks to 9 weeks + 6 days

Exclusion Criteria:

* Pregnant women with singleton or twin pregnancy
* Pregnant women before 6 weeks (higher incidence of spontaneous vanishing twin)
* Pregnant women after 9 weeks + 6 days (the technique is difficult to apply)
* Pelvic or genital infection
* Hemorrhagic blood disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Success of the procedure | 5 minutes after the end of fetal reduction
  Number of gestational sacs in which fetal heart activity will stop

SECONDARY OUTCOMES:
Duration of the fetal reduction procedure | 5 minutes after the end of the procedure when cessation of fetal heart is confirmed
  Duration in minutes needed for each fetus to be reduced (from time of introduction of embryo reduction needle into the gestational sac till fetal heart activity stops)
Post-operative vaginal spotting or bleeding | within the first week of the procedure i.e. from the end of the procedure till 7 days after the procedure
  Number of participants who will develop vaginal spotting or bleeding related to the procedure
Gestational age at birth | On the same day of delivery
  age of pregnancy in weeks and days at time of delivery
Fetal birth weight | On the same day of delivery
  fetal weight in grams at time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Omar, MD, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No